CLINICAL TRIAL: NCT05171465
Title: Intrasaccular neCk Occlusion deVice Treatment of Intracranial Aneurysm in Acute Subarachnoid hemorRhAGE
Acronym: COVERAGE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)564/2021
Record Dates: First submitted 2021-12-10; First posted 2021-12-29 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2021-12

CONDITIONS: Subarachnoid Hemorrhage; Subarachnoid Hemorrhage, Aneurysmal
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Neqstent or Contour — All patients included will be treated the same: after catheterizing the affected vessel and microcatheterizing the aneurysm with a microcatheter of 0.021'' or 0.027'', the intrasaccular device (Neqstent® or Contour®) will be positioned. Depending of the operator preference, the use of an intrasaccular device could be associated with coiling (mandatory in the case of Neqstent®). Treatment must be performed without previous double antiplatelet treatment (allowing antiplatelet after aneurysm exclusion). Before the treatment all patients should undergo a flat panel CT.

SUMMARY:
Rationale: Intrasaccular neck occlusion devices have been used for unruptured aneurysm without safety concerns and good occlusion rates. In the setting of a subarachnoid hemorrhage, they could improve the rate of complete occlusion without safety concerns.

Aim: To explore the safety and efficacy of intrasaccular neck occlusion devices in patients with acute subarachnoid hemorrhage caused by a ruptured saccular aneurysm by a one arm prospective registry.

Study outcome: The primary outcomes is the rate of complete occlusion (Raymond-Roy I) and rebleeding at one year follow-up. The primary safety outcome is rate of rebleeding during the admission.

ELIGIBILITY:
Inclusion Criteria:

* Acute subarachnoid hemorrhage due to an intracranial ruptured aneurysm. Diagnosis must be done with acute CT or MRI.
* Intracranial saccular aneurysm with neck diameter 2-11mm and neck-dome height ≥2 mm.
* Clinical severity measured by World Federation Neurological Surgeons scale score ≤ III.
* Age ≥18 years.
* Previous modified Rankin scale ≤2.
* Informed consent obtained from the patient or acceptable patient surrogate.

Exclusion Criteria:

* Hemodynamically unstable patients with requirement of advanced vital support.
* Patients with limited life expectancy (<6 months) due to terminal disease.
* Previous antiplatelet or anticoagulation treatment.
* Participation in any other clinical trial with a drug or device which could influence the outcome.
* Patients with neurological or psychiatric disease that could undermine future evaluations.
* Lack of availability for 12 months tracing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVERAGE study is a multicentric and international study developed in high volume centers with previous experienced using intrasaccular neck occlusion devices.
  Patients that met all eligibility criteria are considered for enrolment. We include patients with SAH due to a ruptured intracranial saccular aneurysm and mild to moderate clinical symptoms (World Federation Neurological Surgeons ≤ III).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy achieving the lack of rebleeding | 12 months
  Efficacy of the intrasaccular neck occlusion device achieving the lack of rebleeding
Efficacy achieving the complete occlusion | 12 months
  Efficacy of the intrasaccular neck occlusion device achieving the complete occlusion defined as Raymond-Roy scale score of I at 12 months follow-up evaluated by an image central core lab.

SECONDARY OUTCOMES:
Analysis of the primary outcomes in different subgroups | 12 months
  Analysis of the primary outcomes in different subgroups: anterior versus vertebrobasilar circulation, narrow versus wide (≥4mm) neck, aneurysm size (<10mm versus ≥10mm).
Efficacy achieving the complete occlusion at end of treatment | 1 day
  Efficacy of the intrasaccular neck occlusion device achieving the complete occlusion defined as Raymond-Roy scale score of I at end of treatment.
Rate of patients who underwent the study treatment. | 1 days
  Rate of patients who were included in the study and finally underwent the study treatment.
Rate of retreatment | 12 months
  Rate of retreatment needed during the follow-up.
Rate of mortality during admission or follow-up. | 12 months
  Rate of mortality during admission or follow-up.
Functional outcome | 12 months
  Functional outcome at 12 months measured by modified Rankin scale.
Rate of vascular thrombosis or acute stroke. | 12 months
  Rate of vascular thrombosis or acute stroke during follow-up.
Rate of early rebleeding. | 30 days.
  Rate of early rebleeding during the admission.
Rate of complications associated with the procedure. | 1 day
  Rate of complications associated with the procedure.

IPD SHARING:
Plan to Share IPD: Yes
Under reasoned request for metaanalysis or pooled data analysis
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From now to the end of the study
Access Criteria: Under reasoned request for metaanalysis or pooled data analysis

REFERENCES:
- [Background] Molyneux AJ, Kerr RS, Yu LM, Clarke M, Sneade M, Yarnold JA, Sandercock P; International Subarachnoid Aneurysm Trial (ISAT) Collaborative Group. International subarachnoid aneurysm trial (ISAT) of neurosurgical clipping versus endovascular coiling in 2143 patients with ruptured intracranial aneurysms: a randomised comparison of effects on survival, dependency, seizures, rebleeding, subgroups, and aneurysm occlusion. Lancet. 2005 Sep 3-9;366(9488):809-17. doi: 10.1016/S0140-6736(05)67214-5. PMID 16139655
- [Background] Molyneux AJ, Kerr RS, Birks J, Ramzi N, Yarnold J, Sneade M, Rischmiller J; ISAT Collaborators. Risk of recurrent subarachnoid haemorrhage, death, or dependence and standardised mortality ratios after clipping or coiling of an intracranial aneurysm in the International Subarachnoid Aneurysm Trial (ISAT): long-term follow-up. Lancet Neurol. 2009 May;8(5):427-33. doi: 10.1016/S1474-4422(09)70080-8. Epub 2009 Mar 28. PMID 19329361
- [Background] Murayama Y, Nien YL, Duckwiler G, Gobin YP, Jahan R, Frazee J, Martin N, Vinuela F. Guglielmi detachable coil embolization of cerebral aneurysms: 11 years' experience. J Neurosurg. 2003 May;98(5):959-66. doi: 10.3171/jns.2003.98.5.0959. PMID 12744354
- [Background] Raymond J, Guilbert F, Weill A, Georganos SA, Juravsky L, Lambert A, Lamoureux J, Chagnon M, Roy D. Long-term angiographic recurrences after selective endovascular treatment of aneurysms with detachable coils. Stroke. 2003 Jun;34(6):1398-403. doi: 10.1161/01.STR.0000073841.88563.E9. Epub 2003 May 29. PMID 12775880
- [Background] Spetzler RF, McDougall CG, Zabramski JM, Albuquerque FC, Hills NK, Russin JJ, Partovi S, Nakaji P, Wallace RC. The Barrow Ruptured Aneurysm Trial: 6-year results. J Neurosurg. 2015 Sep;123(3):609-17. doi: 10.3171/2014.9.JNS141749. Epub 2015 Jun 26. PMID 26115467
- [Background] Spetzler RF, McDougall CG, Zabramski JM, Albuquerque FC, Hills NK, Nakaji P, Karis JP, Wallace RC. Ten-year analysis of saccular aneurysms in the Barrow Ruptured Aneurysm Trial. J Neurosurg. 2019 Mar 8;132(3):771-776. doi: 10.3171/2018.8.JNS181846. Print 2020 Mar 1. PMID 30849758
- [Background] Campi A, Ramzi N, Molyneux AJ, Summers PE, Kerr RS, Sneade M, Yarnold JA, Rischmiller J, Byrne JV. Retreatment of ruptured cerebral aneurysms in patients randomized by coiling or clipping in the International Subarachnoid Aneurysm Trial (ISAT). Stroke. 2007 May;38(5):1538-44. doi: 10.1161/STROKEAHA.106.466987. Epub 2007 Mar 29. PMID 17395870
- [Background] Youssef PP, Dornbos Iii D, Peterson J, Sweid A, Zakeri A, Nimjee SM, Jabbour P, Arthur AS. Woven EndoBridge (WEB) device in the treatment of ruptured aneurysms. J Neurointerv Surg. 2021 May;13(5):443-446. doi: 10.1136/neurintsurg-2020-016405. Epub 2020 Jul 21. PMID 32719167